CLINICAL TRIAL: NCT04088110
Title: Pyrotinib Maleate Combined With Trastuzumab Plus Aromatase Inhibitor in the First-line Treatment of Advanced HER2-positive/HR-positive Breast Cancer Phase II Study
Brief Title: Pyrotinib Combined With Trastuzumab Plus Aromatase Inhibitor in Treatment of Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Arise-FJ-B102
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer Female; HER2-positive Breast Cancer; Hormone Receptor Positive Malignant Neoplasm of Breast; Metastatic Breast Cancer; Breast Diseases; Hormone Receptor Positive Tumor
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — pyrotinib; Drug Evaluation; Trastuzumab; Aromatase Inhibitors; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib and trastuzumab plus aromatase inhibito (Experimental): Participants will receive pyrotinib in combination with trastuzumab plus AI until pre-defined study end, disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab; Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib were administered 400 mg orally daily. Oral administration within 30 minutes after breakfast, and continuous administration for 21 days for 1 cycle.
  Other Names: Study drug
Drug: Trastuzumab — Trastuzumab were administered every 3 weeks intravenously (8 mg/kg loading doses followed by 6 mg/kg maintenance doses).
  Other Names: Herceptin®
Drug: Aromatase Inhibitors — The investigator chose an aromatase inhibitor (either anastrozole, letrozole or exemestane 1 mg/2.5 mg/25 mg), once daily, oral.
  Other Names: anastrozole, letrozole or exemestane

SUMMARY:
This study is a single-arm, open-label, phase II study, comparing the efficacy and safety of pyrotinib plus trastuzumab and aromatase inhibitors, in the treatment of HR (hormone receptor)+/HER2 (human epidermal growth factor receptor 2) + MBC and inoperable LABC patients.

DETAILED DESCRIPTION:
This is a exploratory, single-arm, open-label,multicenter phase II trial. Our primary purpose is to compare that PFS of patients with pyrotinib plus trastuzumab and AI for HER2-positive and hormone receptor-positive MBC or locally advanced breast cancer (LABC).

In treatment period, patients will be administrated pyrotinib plus trastuzumab and aromatase inhibitors, every 21 days for 1 cycle, until disease progression, toxicity intolerance, withdrawal of informed consent, patients judged must be terminated study termination.

The imaging evaluation was performed according to the RECIST 1.1 criteria every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years,≤70 years, female;
2. Postmenopausal or pre-menopausal with ovarian function suppression;
3. with or without measurable lesion evaluable according to Response Evaluation Criteria In Solid Tumors Version 1.1;
4. Metastatic or inoperable local advanced Invasive breast cancer;
5. HER2-positive breast cancer;
6. HR-positive breast cancer;
7. LVEF ≥55%;QT interva<470 ms;
8. Eastern Cooperative Oncology Group(ECOG) scale 0-1;
9. Life expectancy ≥3 months;

Exclusion Criteria:

1. Previous systemic non-hormonal anticancer therapy in the metastatic or advanced breast cancer setting;
2. Received endocrine therapy within 7 days before randomization;Uncontrolled central nervous system metastases;
3. Disease-free interval from completion of adjuvant/neo-adjuvant systemic non-hormonal treatment to recurrence of within 6 months.
4. Other malignancies within the last 5 years, except for carcinoma in situ of the cervix or basal cell carcinoma.
5. Major surgical procedure or significant traumatic injury within 28 days prior to study treatment start or anticipation of the need for major surgery during the course of study treatment
6. Severe organ dysfunction as assessed by signs and symptoms, laboratory studies and rapid progression of disease, which leading to a clinical indication for chemotherapy.
7. History of CHF of any New York Heart Association (NYHA) criteria, or serious cardiac arrhythmia requiring treatment (exception, atrial fibrillation, paroxysmal supraventricular tachycardia);
8. History of myocardial infarction within 6 months of randomization;
9. History of LVEF decline to below 50% during or after prior trastuzumab neo-adjuvant or adjuvant therapy;
10. Pregnant or lactating women;
11. QT interval>470 ms;
12. Serious concomitant diseases (including severe hypertension, severe diabetes, active infection, thyroid disease, etc.) that are harmful to the patient's safety or affect the patient's completion of the study;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization to 36 month
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
  The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.

SECONDARY OUTCOMES:
Objective Overall Response Rate (ORR) | From randomization to 36 month
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The ORR will be reported by percentage with each arms and appropriate confidence intervals.
Duration of Response (DoR) | From randomization to 36 month
  DoR is defined as date of initial confirmed PR/CR until date of progressive disease or death from any cause. PR or CR or SD is according to RECIST version 1.1.
  The DoR will be estimated using Kaplan-Meier method. Kaplan-Meier curves, median DoR, hazard ratio with appropriate confidence intervals will be reported.
Overall Survival (OS) | From randomization to 36 month
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization.
  The OS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Xi, PhD, Study Chair — Fuzhou General Hospital
Locations (1):
- Fuzhou general hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No